CLINICAL TRIAL: NCT03688165
Title: The Effects of Gait Rehabilitation Using Treadmill-based Robotics (Exoskeletons or End-effectors) Versus Traditional Physical Therapy in Stroke Survivors: a Multicenter Controlled Non-randomized Trial
Brief Title: The Effects of Gait Rehabilitation After Stroke by Treadmill-based Robotics Versus Traditional Gait Training
Acronym: TREAD_STROKE
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Ospedale Santo Stefano (Other); APSS Trento (Unknown); Azienda Sanitaria n. 4 Chiavarese (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Azienda Ospedaliera San Gerardo di Monza (Other); University Hospital of Ferrara (Other); Privatklinik Villa Melitta (Other); Centro Ricerche Cliniche di Verona (Other); Unità di Neuroriabilitazione, HABILITA (Unknown); Istituto Piero Redaelli, Milano (Unknown); S. Anna Hospital (Other); Azienda Sanitaria Locale n.2 Savonese (Other); Fondazione Centri di Riabilitazione Padre Pio Onlus (Unknown); Habilita, Ospedale di Sarnico (Other); I.R.C.C.S. Fondazione Santa Lucia (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Azienda Socio Sanitaria Territoriale di Mantova (Other)
Responsible Party: Sponsor
Other Study IDs: RP 19/17
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Acute Stroke; Chronic Stroke
Keywords: Stroke; End-effector; Exoskeleton; Treadmill-based gait training; Over-ground gait training; Rehabilitation; Functional Gait Recovery; Hemiparesis; Treadmill-based robotic systems
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Treadmill-based Robotic Gait Training: The Treadmill-based Robotic Gait Training (TRGT) period will last 20 sessions, 3-5 days/week for at least 400' of exercise totally. The parameters to be respected for the robotic training will be the following for all patients: 0.9 km / h starting speed up to a maximum of 2.5 km / h; weight support not exceeding 40-45% of the body weight at the beginning and gradual progressive reduction depending on the case; for Lokomat: maximum assistance required at the start of treatment and gradual decrease during the treatment. The TRGT will always be associated with the traditional gait rehabilitation, and will be part of the Individual Rehabilitation Project which normally includes 3 hours of rehabilitation treatments for patients in the subacute phase, 60' of treatment for those in chronic phase.
  Interventions: Device: Treadmill-based Robotic Gait Training
- Traditional Over-ground Gait Training: The Traditional Over-ground Gait Training (TOGT) period will last 20 sessions, 3-5 days / week for a total time that corresponds to the same total time of traditional overground gait training, or at least 400' totally at the end of the period.
  By Traditional Therapy we mean any technical approach aimed at achieving control of the postural passages from sitting upright, of load transfer in laterality and antero-posterior in orthostatism and reorganization of the step up to the assisted path to the parallels and then with various aids.
  Interventions: Other: Traditional Over-ground Gait Training

INTERVENTIONS:
Device: Treadmill-based Robotic Gait Training — All the stroke survivors admitted to the participating centers and eligible for the study will follow a gait training protocol (treadmill-based or overground). The data will be registered at baseline (T0), end of treatment (T1) and at three months follow up (T2). All robotic systems used for the study (Lokomat Pro - Hocoma AG, Volketswil, Switzerland); G-EO System - Reha technologies, Italy) are treadmill-based and do not provide the over-ground gait training. They are characterized by the possibility of a programmable weight support, as well as speed and stride length. The data relating to the patients' training is always displayed and stored with a computerized control system.
  Other Names: Over-ground Traditional Gait Training
  Groups: Treadmill-based Robotic Gait Training
Other: Traditional Over-ground Gait Training — Traditional treatment for gait training consists in any conventional technical approach aimed at achieving control of the postural passages from sitting upright, of load transfer in laterality and antero-posterior in orthostatism and reorganization of the step up to the assisted path to the parallels and then with various aids.
  Groups: Traditional Over-ground Gait Training

SUMMARY:
This multicenter non-randomized controlled trial aims to investigate the effectiveness (an increase of the walking speed in the 10 Meter Walk Test - 10MWT) of the robotic treatment with exoskeleton or end-effector system compared to the conventional rehabilitative treatment for the gait recovery after stroke, and to compare the possible different efficacy of end-effector and exoskeleton systems in the various post-stroke disability frameworks.

All the eligible subjects admitted to rehabilitation centers, both in the subacute phase will be recorded. The experimental group will follow a set of robotic gait training on stationary robotic systems which do not provide overground gait training (Lokomat Pro - Hocoma AG, Volketswil, Switzerland; G-EO System - Reha technologies, Italy). While, the control group will follow traditional gait training composed of all those exercises which promote the recovery of walking ability (please, see the details of the interventions).

DETAILED DESCRIPTION:
This multicenter non-randomized controlled trial aims:

* to investigate the efficacy of a treadmill-based robotic treatment (both end-effector and exoskeleton) compared to the conventional rehabilitative treatment on gait recovery in stroke survivors;
* to verify different effects of the end-effector or exoskeleton system on stroke subjects with different disabilities.

All the eligible subjects (please, see the inclusion and exclusion criteria), admitted to the study participant centers for rehabilitation treatment, will be recorded at any stage of the rehabilitation program (subacute or chronic phase).

The patient's recruitment will run following the authorization of the respective Ethics Committees for 12 months.

Both experimental or control group will be undergone to 20 sessions of treatments, from 3 to 5 times per week, each lasting 60 minutes ( for a total of 400 minutes of treatment) All robotic systems used in this study for the experimental group (Lokomat Pro - Hocoma AG, Volketswil, Switzerland; G-EO System - Rehatechnologies, Italy) are treadmill-based and do not provide the over-ground gait training. They are characterized by the possibility of a programmable load suspension, as well as speed, stride length. The patient's activity with the related data is always displayed and stored with a computerized control system.

The control group will follow a traditional gait rehabilitation for the same duration as the experimental group.

The clinical assessments and data analysis will be carried out blindly.

ELIGIBILITY:
Inclusion Criteria:

* age ≤ 85 years;
* first ever event of pyramidal hemisyndrome (any functional level and etiology);
* possibility to understand and execute simple instructions, for performing correctly the robot exercise;
* for chronic patients: Functional Ambulation Category (FAC)> 1.

Exclusion Criteria:

* bilateral impairment;
* Walking Handicap Scale (WHS) <5 before the acute event;
* cognitive or behavioral deficit as to compromise the comprehension of the robotic training;
* neurolytic treatment with botulinum toxin in the previous 3 months and/or during the study (including follow up);
* use of other technologies (robots, FES, TDCS ...) during the study;
* impossibility or non-availability to provide the informed consent;
* cardiorespiratory gravity-morbidity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the subjects admitted to the participating centers for rehabilitation treatment following a first ever stroke, both in subacute or chronic phase.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in 10 Meter Walk Test (10MWT) | at baseline (T0), at 2 months-the end of treatment (T1) and at 3 months after the end of rehabilitation-follow up (T2)
  This test will assess the patient's speed during gait. Patients will be asked to walk at their preferred maximum and safe speed. Patients will be positioned 1 meter before the start line and instructed to walk 10 meters, and pass the end line approximately 1 meter after. The distance before and after the course are meant to minimize the effect of acceleration and deceleration. Time will be measured using a stopwatch and recorded to the one hundredth of a second (ex: 2.15 s). The test will be recorded 3 times, with adequate rests between them. The average of the 3 times should be recorded.

SECONDARY OUTCOMES:
Change in Timed Up and Go test (TUG) | at baseline (T0), at 2 months-the end of treatment (T1) and at 3 months after the end of rehabilitation-follow up (T2)
  The TUG is a test used to assess mobility, balance, and walking in people with balance impairments. The subject must stand up from a chair (which should not be leant against a wall), walk a distance of 3 meters, turn around, walk back to the chair and sit down - all performed as quickly and as safely as possible. Time will be measured using a chronometer.
Change in 6 Minute Walking Test (6MWT) | at baseline (T0), at 2 months-the end of treatment (T1) and at 3 months after the end of rehabilitation-follow up (T2)
  The 6MWT measures the distance a subject covers during an indoor gait on a flat, hard surface in 6 minutes, using assistive devices, as necessary. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The minimal detectable change in distance for people with sub-acute stroke is 60.98 meters. The 6MWT is a patient self-paced walk test and assesses the level of functional capacity. Patients are allowed to stop and rest during the test. However, the timer does not stop. If the patient is unable to complete the test, the time is stopped at that moment. The missing time and the reason of the stop are recorded. This test will be administered while wearing a pulse oximeter to monitor heart rate and oxygen saturation, also integrated with Borg scale to assess dyspnea.
Change in Trunk Control Test (TCT) | at baseline (T0), at 2 months-the end of treatment (T1) and at 3 months after the end of rehabilitation-follow up (T2)
  The TCT assesses the motor impairment in stroke patients and it's correlated with eventual walking ability. Testing is done with the patient lying on a bed: (1) roll to weak side. (2) roll to strong side. (3) balance in sitting position on the edge of the bed with the feet off the ground for at least 30. (4) sit up from lying down. Total score: 0-100.
Change in Motricity Index (MI) | at baseline (T0), at 2 months-the end of treatment (T1) and at 3 months after the end of rehabilitation-follow up (T2)
  The MI aims to evaluate lower limb motor impairment after stroke, administrated on both sides.
  Items to assess the lower limbs are 3, scoring from 0 to 33 each: (1) ankle dorsiflexion with foot in a plantar flexed position (2) knee extension with the foot unsupported and the knee at 90° (3) hip flexion with the hip at 90° moving the knee as close as possible to the chin. (no movement: 0, palpable flicker but no movement: 9, movement but not against gravity :14, movement against gravity movement against gravity: 19, movement against resistance: 25, normal:33)
  1 leg score for each side = SUM (points for the 3 leg tests) + 1 Interpretation: minimum score: 0; maximum score:100
Change in ModifiedAshworth Scale (MAS) | at baseline (T0), at 2 months-the end of treatment (T1) and at 3 months after the end of rehabilitation-follow up (T2)
  The MAS is a 6 point ordinal scale used for grading hypertonia in individuals with neurological diagnoses. A score of 0 on the scale indicates no increase in tone while a score of 4 indicates rigidity. Tone is scored by passively moving the individual's limb and assessing the amount of resistance to movement felt by the examiner.
Change in Modified Barthel Index (mBI) | at baseline (T0), at 2 months-the end of treatment (T1) and at 3 months after the end of rehabilitation-follow up (T2)
  To assess the level of disability during the indoor and outdoor activities of daily living
Change in Walking Handicap Scale (WHS) | at baseline (T0), at 2 months-the end of treatment (T1) and at 3 months after the end of rehabilitation-follow up (T2)
  WHS is a classification of 6 functional walking categories, considered as a participation category of the ICF because of its 3 items referred to community ambulation.

OTHER OUTCOMES:
Functional Ambulation Category (FAC) | at baseline (T0) only
  FAC is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Franceschini, MD, Study Chair — IRCCS San Raffaele Pisana; Sanaz Pournajaf, Dr, Principal Investigator — IRCCS San Raffaele Pisana
Locations (4):
- Italy (4):
  - IRCCS San Raffaele Pisana, Roma, Italy
  - U.O.C. Medicina Fisica e Riabilitazione, osp.S.Gerardo, Monza, Lombardy
  - Irccs Centro Neurolesi Bonino Pulejo, Messina
  - Irccs Fondazione Santa Lucia, Roma

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcome measures, including assessment results and relevant demographic data, can be shared in compliance with ethical and legal requirements upon specific request to the Study PI.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting information are available upon request starting from the official publication date and will remain accessible for a period of two years after study completion.
Access Criteria: Access will be granted upon specific request to the Principal Investigator, Study Chair, or designated central study contact. Researchers must submit a formal proposal outlining the intended use of the data, which will be reviewed for scientific merit and ethical compliance. Approved requests will receive access through a secure data-sharing platform.
URL: https://www.mdpi.com/2077-0383/12/2/439

REFERENCES:
- [Background] Awad LN, Reisman DS, Pohlig RT, Binder-Macleod SA. Identifying candidates for targeted gait rehabilitation after stroke: better prediction through biomechanics-informed characterization. J Neuroeng Rehabil. 2016 Sep 23;13(1):84. doi: 10.1186/s12984-016-0188-8. PMID 27663199
- [Background] Bae YH, Ko YJ, Chang WH, Lee JH, Lee KB, Park YJ, Ha HG, Kim YH. Effects of Robot-assisted Gait Training Combined with Functional Electrical Stimulation on Recovery of Locomotor Mobility in Chronic Stroke Patients: A Randomized Controlled Trial. J Phys Ther Sci. 2014 Dec;26(12):1949-53. doi: 10.1589/jpts.26.1949. Epub 2014 Dec 25. PMID 25540505
- [Background] Balami JS, Buchan AM. Complications of intracerebral haemorrhage. Lancet Neurol. 2012 Jan;11(1):101-18. doi: 10.1016/S1474-4422(11)70264-2. PMID 22172625
- [Background] Bejot Y, Daubail B, Giroud M. Epidemiology of stroke and transient ischemic attacks: Current knowledge and perspectives. Rev Neurol (Paris). 2016 Jan;172(1):59-68. doi: 10.1016/j.neurol.2015.07.013. Epub 2015 Dec 21. PMID 26718592
- [Background] Blackburn M, van Vliet P, Mockett SP. Reliability of measurements obtained with the modified Ashworth scale in the lower extremities of people with stroke. Phys Ther. 2002 Jan;82(1):25-34. doi: 10.1093/ptj/82.1.25. PMID 11784275
- [Background] Bohannon RW, Andrews AW, Glenney SS. Minimal clinically important difference for comfortable speed as a measure of gait performance in patients undergoing inpatient rehabilitation after stroke. J Phys Ther Sci. 2013 Oct;25(10):1223-5. doi: 10.1589/jpts.25.1223. Epub 2013 Nov 20. PMID 24259762
- [Background] Bowden MG, Balasubramanian CK, Behrman AL, Kautz SA. Validation of a speed-based classification system using quantitative measures of walking performance poststroke. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):672-5. doi: 10.1177/1545968308318837. PMID 18971382
- [Background] Chang WH, Kim YH. Robot-assisted Therapy in Stroke Rehabilitation. J Stroke. 2013 Sep;15(3):174-81. doi: 10.5853/jos.2013.15.3.174. Epub 2013 Sep 27. PMID 24396811
- [Background] Chollet F, Albucher JF. Strategies to augment recovery after stroke. Curr Treat Options Neurol. 2012 Dec;14(6):531-40. doi: 10.1007/s11940-012-0196-3. PMID 22865294
- [Background] Danzl MM, Chelette KC, Lee K, Lykins D, Sawaki L. Brain stimulation paired with novel locomotor training with robotic gait orthosis in chronic stroke: a feasibility study. NeuroRehabilitation. 2013;33(1):67-76. doi: 10.3233/NRE-130929. PMID 23949035
- [Background] Demeurisse G, Demol O, Robaye E. Motor evaluation in vascular hemiplegia. Eur Neurol. 1980;19(6):382-9. doi: 10.1159/000115178. PMID 7439211
- [Background] Dobkin BH. Clinical practice. Rehabilitation after stroke. N Engl J Med. 2005 Apr 21;352(16):1677-84. doi: 10.1056/NEJMcp043511. PMID 15843670
- [Background] Fulk GD, Echternach JL. Test-retest reliability and minimal detectable change of gait speed in individuals undergoing rehabilitation after stroke. J Neurol Phys Ther. 2008 Mar;32(1):8-13. doi: 10.1097/NPT0b013e31816593c0. PMID 18463550
- [Background] Hesse S, Uhlenbrock D, Werner C, Bardeleben A. A mechanized gait trainer for restoring gait in nonambulatory subjects. Arch Phys Med Rehabil. 2000 Sep;81(9):1158-61. doi: 10.1053/apmr.2000.6280. PMID 10987154
- [Background] Hesse S, Waldner A, Tomelleri C. Innovative gait robot for the repetitive practice of floor walking and stair climbing up and down in stroke patients. J Neuroeng Rehabil. 2010 Jun 28;7:30. doi: 10.1186/1743-0003-7-30. PMID 20584307
- [Background] Hesse S, Schattat N, Mehrholz J, Werner C. Evidence of end-effector based gait machines in gait rehabilitation after CNS lesion. NeuroRehabilitation. 2013;33(1):77-84. doi: 10.3233/NRE-130930. PMID 23949037
- [Background] Hidler JM, Wall AE. Alterations in muscle activation patterns during robotic-assisted walking. Clin Biomech (Bristol). 2005 Feb;20(2):184-93. doi: 10.1016/j.clinbiomech.2004.09.016. PMID 15621324
- [Background] Hornby TG, Campbell DD, Kahn JH, Demott T, Moore JL, Roth HR. Enhanced gait-related improvements after therapist- versus robotic-assisted locomotor training in subjects with chronic stroke: a randomized controlled study. Stroke. 2008 Jun;39(6):1786-92. doi: 10.1161/STROKEAHA.107.504779. Epub 2008 May 8. PMID 18467648
- [Background] Kelley CP, Childress J, Boake C, Noser EA. Over-ground and robotic-assisted locomotor training in adults with chronic stroke: a blinded randomized clinical trial. Disabil Rehabil Assist Technol. 2013 Mar;8(2):161-8. doi: 10.3109/17483107.2012.714052. Epub 2012 Sep 20. PMID 22992166
- [Background] Kolominsky-Rabas PL, Weber M, Gefeller O, Neundoerfer B, Heuschmann PU. Epidemiology of ischemic stroke subtypes according to TOAST criteria: incidence, recurrence, and long-term survival in ischemic stroke subtypes: a population-based study. Stroke. 2001 Dec 1;32(12):2735-40. doi: 10.1161/hs1201.100209. PMID 11739965
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Lee IW, Kim YN, Lee DK. Effect of a virtual reality exercise program accompanied by cognitive tasks on the balance and gait of stroke patients. J Phys Ther Sci. 2015 Jul;27(7):2175-7. doi: 10.1589/jpts.27.2175. Epub 2015 Jul 22. PMID 26311949
- [Background] Mazzoleni S, Focacci A, Franceschini M, Waldner A, Spagnuolo C, Battini E, Bonaiuti D. Robot-assisted end-effector-based gait training in chronic stroke patients: A multicentric uncontrolled observational retrospective clinical study. NeuroRehabilitation. 2017;40(4):483-492. doi: 10.3233/NRE-161435. PMID 28211822
- [Background] Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1314-9. doi: 10.1016/j.apmr.2007.06.764. PMID 17908575
- [Background] Mehrholz J, Thomas S, Werner C, Kugler J, Pohl M, Elsner B. Electromechanical-assisted training for walking after stroke. Cochrane Database Syst Rev. 2017 May 10;5(5):CD006185. doi: 10.1002/14651858.CD006185.pub4. PMID 28488268
- [Background] Moreland JD, Depaul VG, Dehueck AL, Pagliuso SA, Yip DW, Pollock BJ, Wilkins S. Needs assessment of individuals with stroke after discharge from hospital stratified by acute Functional Independence Measure score. Disabil Rehabil. 2009;31(26):2185-95. doi: 10.3109/09638280902951846. PMID 19903128
- [Background] Ochi M, Wada F, Saeki S, Hachisuka K. Gait training in subacute non-ambulatory stroke patients using a full weight-bearing gait-assistance robot: A prospective, randomized, open, blinded-endpoint trial. J Neurol Sci. 2015;353(1-2):130-6. doi: 10.1016/j.jns.2015.04.033. Epub 2015 May 1. PMID 25956233
- [Background] Paolucci S, Bragoni M, Coiro P, De Angelis D, Fusco FR, Morelli D, Venturiero V, Pratesi L. Quantification of the probability of reaching mobility independence at discharge from a rehabilitation hospital in nonwalking early ischemic stroke patients: a multivariate study. Cerebrovasc Dis. 2008;26(1):16-22. doi: 10.1159/000135648. Epub 2008 May 30. PMID 18511867
- [Background] Perry J, Garrett M, Gronley JK, Mulroy SJ. Classification of walking handicap in the stroke population. Stroke. 1995 Jun;26(6):982-9. doi: 10.1161/01.str.26.6.982. PMID 7762050
- [Background] Peurala SH, Tarkka IM, Pitkanen K, Sivenius J. The effectiveness of body weight-supported gait training and floor walking in patients with chronic stroke. Arch Phys Med Rehabil. 2005 Aug;86(8):1557-64. doi: 10.1016/j.apmr.2005.02.005. PMID 16084808
- [Background] Picelli A, Chemello E, Castellazzi P, Roncari L, Waldner A, Saltuari L, Smania N. Combined effects of transcranial direct current stimulation (tDCS) and transcutaneous spinal direct current stimulation (tsDCS) on robot-assisted gait training in patients with chronic stroke: A pilot, double blind, randomized controlled trial. Restor Neurol Neurosci. 2015;33(3):357-68. doi: 10.3233/RNN-140474. PMID 26410579
- [Background] Rand D, Eng JJ, Liu-Ambrose T, Tawashy AE. Feasibility of a 6-month exercise and recreation program to improve executive functioning and memory in individuals with chronic stroke. Neurorehabil Neural Repair. 2010 Oct;24(8):722-9. doi: 10.1177/1545968310368684. Epub 2010 May 11. PMID 20460494
- [Background] Rosa MC, Marques A, Demain S, Metcalf CD. Fast gait speed and self-perceived balance as valid predictors and discriminators of independent community walking at 6 months post-stroke--a preliminary study. Disabil Rehabil. 2015;37(2):129-34. doi: 10.3109/09638288.2014.911969. Epub 2014 Apr 23. PMID 24754638
- [Background] Sale P, Franceschini M, Waldner A, Hesse S. Use of the robot assisted gait therapy in rehabilitation of patients with stroke and spinal cord injury. Eur J Phys Rehabil Med. 2012 Mar;48(1):111-21. PMID 22543557
- [Background] Schwartz I, Meiner Z. Robotic-assisted gait training in neurological patients: who may benefit? Ann Biomed Eng. 2015 May;43(5):1260-9. doi: 10.1007/s10439-015-1283-x. Epub 2015 Feb 28. PMID 25724733
- [Background] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Background] Swinnen E, Baeyens JP, Knaepen K, Michielsen M, Hens G, Clijsen R, Goossens M, Buyl R, Meeusen R, Kerckhofs E. Walking with robot assistance: the influence of body weight support on the trunk and pelvis kinematics. Disabil Rehabil Assist Technol. 2015 May;10(3):252-7. doi: 10.3109/17483107.2014.888487. Epub 2014 Feb 11. PMID 24512196
- [Background] Taqi MA, Vora N, Callison RC, Lin R, Wolfe TJ. Past, present, and future of endovascular stroke therapies. Neurology. 2012 Sep 25;79(13 Suppl 1):S213-20. doi: 10.1212/WNL.0b013e31826959e5. PMID 23008401
- [Background] Taveggia G, Borboni A, Mule C, Villafane JH, Negrini S. Conflicting results of robot-assisted versus usual gait training during postacute rehabilitation of stroke patients: a randomized clinical trial. Int J Rehabil Res. 2016 Mar;39(1):29-35. doi: 10.1097/MRR.0000000000000137. PMID 26512928
- [Background] Thrift AG, Srikanth VK, Nelson MR, Kim J, Fitzgerald SM, Gerraty RP, Bladin CF, Phan TG, Cadilhac DA. Risk factor management in survivors of stroke: a double-blind, cluster-randomized, controlled trial. Int J Stroke. 2014 Jul;9(5):652-7. doi: 10.1111/j.1747-4949.2012.00933.x. Epub 2012 Dec 11. PMID 23231528
- [Background] Tong RK, Ng MF, Li LS. Effectiveness of gait training using an electromechanical gait trainer, with and without functional electric stimulation, in subacute stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2006 Oct;87(10):1298-304. doi: 10.1016/j.apmr.2006.06.016. PMID 17023237
- [Background] Vahlberg B, Cederholm T, Lindmark B, Zetterberg L, Hellstrom K. Factors related to performance-based mobility and self-reported physical activity in individuals 1-3 years after stroke: a cross-sectional cohort study. J Stroke Cerebrovasc Dis. 2013 Nov;22(8):e426-34. doi: 10.1016/j.jstrokecerebrovasdis.2013.04.028. Epub 2013 May 28. PMID 23721615
- [Background] van de Port IG, Kwakkel G, Lindeman E. Community ambulation in patients with chronic stroke: how is it related to gait speed? J Rehabil Med. 2008 Jan;40(1):23-7. doi: 10.2340/16501977-0114. PMID 18176733
- [Background] van Hedel HJ, Wirz M, Dietz V. Assessing walking ability in subjects with spinal cord injury: validity and reliability of 3 walking tests. Arch Phys Med Rehabil. 2005 Feb;86(2):190-6. doi: 10.1016/j.apmr.2004.02.010. PMID 15706542
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Waldner A, Tomelleri C, Hesse S. Transfer of scientific concepts to clinical practice: recent robot-assisted training studies. Funct Neurol. 2009 Oct-Dec;24(4):173-7. PMID 20412721
- [Background] Zhang X, Yue Z, Wang J. Robotics in Lower-Limb Rehabilitation after Stroke. Behav Neurol. 2017;2017:3731802. doi: 10.1155/2017/3731802. Epub 2017 Jun 8. PMID 28659660